CLINICAL TRIAL: NCT07156981
Title: Investigation of Effects of Physiotherapy in Children With Hirschsprung's Disease
Brief Title: Effects of Physiotherapy in Children With Hirschsprung's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, Professor, Ankara Yildirim Beyazıt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TABED1/1561/2025
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hirschsprung Disease
MeSH Terms: conditions — Hirschsprung Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy (Other): Physiotherapy program will be performed
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Physiotherapy — The treatment program will include patient education, lifestyle recommendations, breathing exercises, pelvic floor muscle training, and stabilization exercises. The treatment program will last for a total of 8 weeks.

SUMMARY:
The aim of our study is to investigate the effects of physiotherapy in children with Hirschsprung's disease who have bowel symptoms after surgery.

DETAILED DESCRIPTION:
Hirschsprung's disease is a developmental disorder of the enteric nervous system characterized by the absence of ganglion cells in the distal intestine, resulting in functional intestinal obstruction. The treatment applied after diagnosis is surgical. Although individuals with a history of surgery due to Hirschsprung's disease generally have normal bowel and urinary function, it has been reported that they have a higher prevalence of fecal incontinence and constipation and a lower quality of life related to the gastrointestinal system. However, there are few studies evaluating the use of physiotherapy in the management of postoperative bowel symptoms in children with Hirschsprung's disease.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-18 who have undergone surgery for Hirschsprung's disease and have intestinal symptoms, and who come for routine check-ups.
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of a congenital and/or chronic disease
* Those with missing assessment parameters
* Having a history of any additional orthopedic, neurological or psychiatric disease that will affect the evaluation parameters
* Loss of sensation
* Mental retardation

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Bowel function | before and after treatment (8-week change)
  Bowel function will be evaluated with a bowel diary. They will be asked to keep a bowel diary for 1 week, including the number and type of daily stools and the number of incontinent stools.

SECONDARY OUTCOMES:
Constipation | before and after treatment (8-week change)
  Children's constipation will be evaluated with the Rome IV criteria. These criteria include; two or less defecation per week, fecal incontinence at least once a week, history of holding/ delaying the large toilet, painful and difficult bowel movements, presence of large feces in the rectum, presence of a history of large feces that can block the toilet. An increase in the number of symptoms indicates the severity of constipation.
Pelvic floor muscle function | before and after treatment (8-week change)
  Pelvic floor muscle function will be evaluated with palpation form anus. The presence of correct contraction and relaxation of the pelvic floor muscle will be determined.
Life quality | before and after treatment (8-week change)
  Life quality will be assessed with the Pediatric Quality of Life Inventory (PedsQL). The PedsQL consists of 23 items. It are scored between 0-100. The higher the total score of the life quality, the better health-related life quality is perceived.
Perception of improvement | after treatment (8-week change)
  Subjective perception of improvement will be assessed as -1 (worse), 0 (no change) and 1 (better).
Compliance with recommendations | after treatment (8-week change)
  Compliance with post-treatment recommendations will be assessed with the Visual Analog Scale (VAS). The VAS is a horizontal line with "0" at one end as "never compliance" and '10' at the other end as "always compliance".

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University